CLINICAL TRIAL: NCT03854578
Title: A Single Dose, Randomized, Placebo Controlled Phase I Study on the Effects of BI 1358894 on Functional MRI Measurements in an Emotional Processing Paradigm in Patients With Major Depressive Disorder
Brief Title: A Study in People With Depression to Test the Effects of BI 1358894 on Parts of the Brain That Are Involved in Emotions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1402-0003; 2017-004763-12 (EudraCT Number)
Record Dates: First submitted 2019-02-25; First posted 2019-02-26 (Actual); Results first posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Depressive Disorder, Major
MeSH Terms: conditions — Depressive Disorder, Major | interventions — TRPC inhibitor BI 1358894; Citalopram

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- BI 1358894 (Experimental)
  Interventions: Drug: BI 1358894
- Citalopram (Experimental)
  Interventions: Drug: Citalopram
- Placebo matching BI 1358894 (Experimental)
  Interventions: Drug: Placebo matching BI 1358894

INTERVENTIONS:
Drug: BI 1358894 — Film-coated tablet
  Arms: BI 1358894
Drug: Placebo matching BI 1358894 — Film-coated tablet
  Arms: Placebo matching BI 1358894
Drug: Citalopram — Film-coated tablet
  Arms: Citalopram

SUMMARY:
To assess the effect of a single dose of BI 1358894 compared to placebo on BOLD responses in modulating brain processing of emotional and cognitive stimuli on the amygdala and related brain structure using fMRI in in unmedicated patients with depression.

ELIGIBILITY:
Inclusion Criteria:

* Patients having a diagnosis of a MDD according to Diagnostic and Statistical Manual of Mental Disorders-V (DSM-V) (single episode or recurrent) with a MADRS total score between ≥ 7 and < 26 at screening.
* Male or female aged 18 to 45 years, inclusive at screening.
* Male or female patients. Women of childbearing potential (WOCBP) and men able to father a child must be ready and able to use highly effective methods of birth control.
* Patients must be, in the opinion of the Investigator, capable of and eligible for completing the fMRI and tasks.
* Patients must be right-handed.
* Patients must have acceptable weight as defined by BMI (weight [kg]/height [m]²) range of 18 to 30 kg/m², inclusive at Visit 1.
* Patients must be a non-smoker or light smoker (≤ 5 cigarettes per day).
* Patients must have signed the informed consent form prior to the first study-related procedure indicating they understand the purpose of and procedures required for the study and are willing to participate in the study.
* Further inclusion criteria apply

Exclusion Criteria:

* Meeting any diagnostic criteria for a major psychiatric disorder (other than MDD), as determined by DSM-V at screening.
* Has received a prescribed medication (including antidepressants) within 28 days prior to Visit 1 (apart from the contraceptive pill) or having received over the counter medication (including pain killers) within 10 days prior to screening. Participants who have taken prescription medication may still be entered into the study, if, in the opinion of the Investigator, the medication received will not interfere with the study procedures or compromise safety.
* Patients where it is foreseen (per investigator judgement) that a delay of initiation of standard of care therapy for the depressive disorder to 14 days after day 1 of Visit 2 is medically not justifiable.
* A history of alcohol or substance dependence or abuse within the last 12 months from Visit 1.
* Has a current or recent history of clinically significant suicidal ideation within the past 6 months, corresponding to a score of 4 or 5 for ideation on the C-SSRS, or a history of suicidal behavior within the past year, as validated by the C-SSRS at screening or treatment visit.
* Has a history of, or presents (in the opinion of the Investigator) with, significant neurological or psychiatric conditions (such as stroke, traumatic brain injury, seizures, space occupying lesions, multiple sclerosis, Parkinson's disease, vascular dementia, transient ischemic attack, schizophrenia, blackouts requiring hospitalisation).
* A planned medical treatment within the study period that might interfere with the study procedures.
* Further exclusion criteria apply

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 73 (Actual)
Dates: Start 2019-03-12 (Actual); Primary Completion 2019-08-27 (Actual); Study Completion 2019-09-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Charité - Universitätsmedizin Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder;
  2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials;
  3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- [Derived] Grimm S, Keicher C, Paret C, Niedtfeld I, Beckmann C, Mennes M, Just S, Sharma V, Fuertig R, Herich L, Mack S, Thamer C, Schultheis C, Weigand A, Schmahl C, Wunder A. The effects of transient receptor potential cation channel inhibition by BI 1358894 on cortico-limbic brain reactivity to negative emotional stimuli in major depressive disorder. Eur Neuropsychopharmacol. 2022 Dec;65:44-51. doi: 10.1016/j.euroneuro.2022.10.009. Epub 2022 Nov 4. PMID 36343427

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A single dose, randomized, placebo controlled Phase I study on the effects of BI 1358894 on functional magnetic resonance Imaging measurements in an emotional processing paradigm in patients with Major Depressive Disorder
Pre-assignment Details: All subjects were screened for eligibility to participate in trial. Subjects visited specialist site to ensure that they met all implemented inclusion/exclusion criteria, Subjects were not to be randomised to trial drug if any of the specific entry criteria was violated
Groups:
- Placebo Matching to BI 1358894: Oral administration of single dose of BI 1358894 matching placebo (4 film-coated tablets) with 240 milliliter (mL) of water after an high-fat, high-calorie breakfast.
  Three hours after the administration of BI 1358894 matching placebo the patient receive 1 film-coated tablet of Placebo.
- Citalopram: Oral administration of single dose of BI 1358894 matching placebo (4 film-coated tablets) with 240 milliliter (mL) of water after an high-fat, high-calorie breakfast.
  Three hours after the first administration of BI 1358894 matching placebo the patient receive a oral administration of single dose of 20 milligram (mg) Citalopram (1 tablet of 20 mg).
- BI 1358894: Oral administration of single dose of 100 milligram (mg) BI 1358894 (4 film-coated tablets of 25 mg) with 240 milliliter (mL) of water after an high-fat, high-calorie breakfast.
  Three hours after the administration of BI 1358894 the patient receive 1 film-coated tablet of Placebo.
Period: Overall Study
Arm/Group | Placebo Matching to BI 1358894 | Citalopram | BI 1358894
Started | 24 | 24 | 25
Completed | 24 | 24 | 25
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Randomised Set (RS): This patient set included all patients who were randomised to receive BI 1358894, Citalopram or placebo. Patients without any post-randomisation data were excluded from the primary and secondary pharmacodynamic analyses
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Matching to BI 1358894 | Citalopram | BI 1358894 | Total
Number analyzed (Participants) | 24 | 24 | 25 | 73
Age, Continuous [Mean (Standard Deviation); unit: Years] | 30.1 (5.6) | 30.8 (6.5) | 31.5 (6.8) | 30.8 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 16 | 13 | 48
  Male | 5 | 8 | 12 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 0 | 2
  Not Hispanic or Latino | 22 | 24 | 25 | 71
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 2 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 1
  White | 23 | 21 | 25 | 69
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Blood Oxygenation Level Depend (BOLD) Signal % Change in an Emotional Paradigm, Based on the Emotional Faces From the Warsaw Set of Emotional Facial Expression Pictures (WSEFEP)
Description: The primary endpoint was the mean BOLD signal % change in an emotional paradigm, based on the emotional faces from the Warsaw Set of Emotional Facial Expression Pictures (WSEFEP) in the corticolimbic system comprising the following eight brain regions of interest:
  * Amygdala left
  * Amygdala right
  * Dorsolateral prefrontal cortex left
  * Dorsolateral prefrontal cortex right
  * Insula left
  * Insula right
  * Anterior cingulate cortex left
  * Anterior cingulate cortex right
Time Frame: A 50 min scan, 6 hours following drug intake.
Population: Evaluable set (ES): This patient set included all randomised patients who performed the functional Magnetic Resonance Imaging (fMRI) measurements and did not experience severe headaches directly before or during the fMRI measurements. In particular, patients who had to be replaced due to severe headaches were excluded from the ES.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Placebo Matching to BI 1358894 | Citalopram | BI 1358894
Number analyzed (Participants) | 24 | 23 | 22
Percent change
  Amygdala left | 0.305 (0.119) | 0.290 (0.134) | 0.223 (0.093)
  Amygdala right | 0.364 (0.136) | 0.291 (0.146) | 0.282 (0.071)
  Dorsolateral prefrontal cortex left | 0.065 (0.146) | 0.044 (0.111) | 0.049 (0.109)
  Dorsolateral prefrontal cortex right | 0.131 (0.202) | 0.117 (0.183) | 0.125 (0.105)
  Insula left | 0.162 (0.146) | 0.110 (0.107) | 0.075 (0.126)
  Insula right | 0.157 (0.133) | 0.137 (0.107) | 0.1205 (0.125)
  Anterior cingulate cortex left | 0.003 (0.121) | -0.027 (0.074) | -0.024 (0.085)
  Anterior cingulate cortex right | -0.008 (0.131) | -0.026 (0.087) | -0.018 (0.101)
Statistical Analysis 1: Comparison: Placebo Matching to BI 1358894 vs BI 1358894; Mean BOLD signal % change/ Amygdala Left; Test type: Other — ANOVA model with treatment (BI 1358894 versus placebo) and severity of depression (MontgomeryÅsberg Depression Rating Scale (MADRS) ≥20 versus <20) as fixed effects. The Citalopram treatment arm was used as a positive control group. It was not planned to compare pharmacodynamic effects between Citalopram and BI 1358894; p = 0.0105, ANOVA; Mean change = -0.08, 90% CI 2-sided [-0.14 to -0.03], Standard Error of Mean 0.03 — Mean change calculated as: BI - Placebo
Statistical Analysis 2: Comparison: Placebo Matching to BI 1358894 vs BI 1358894; Mean BOLD signal % change/ Amygdala Right; Test type: Other — ANOVA model with treatment (BI 1358894 versus placebo) and severity of depression (MADRS ≥20 versus <20) as fixed effects. The Citalopram treatment arm was used as a positive control group. It was not planned to compare pharmacodynamic effects between Citalopram and BI 1358894; p = 0.0134, ANOVA; Mean change = -0.08, 90% CI 2-sided [-0.14 to -0.03], Standard Error of Mean 0.03 — Mean change calculated as: BI - Placebo
Statistical Analysis 3: Comparison: Placebo Matching to BI 1358894 vs BI 1358894; Mean BOLD signal % change/ Anterior Cingulate Cortex Left; Test type: Other — [test comment as in outcome 1, analysis 2]; p = 0.3495, ANOVA; Mean change = -0.03, 90% CI 2-sided [-0.08 to 0.02], Standard Error of Mean 0.03 — Mean change calculated as: BI - Placebo
Statistical Analysis 4: Comparison: Placebo Matching to BI 1358894 vs BI 1358894; Mean BOLD signal % change/ Anterior Cingulate Cortex right; Test type: Other — [test comment as in outcome 1, analysis 2]; p = 0.7008, ANOVA; Mean change = -0.01, 90% CI 2-sided [-0.07 to 0.04], Standard Error of Mean 0.03 — Mean change calculated as: BI - Placebo
Statistical Analysis 5: Comparison: Placebo Matching to BI 1358894 vs BI 1358894; Mean BOLD signal % change/ Dorsolateral Prefrontal Cortex Left; Test type: Other — [test comment as in outcome 1, analysis 2]; p = 0.6635, ANOVA; Mean change = -0.02, 90% CI 2-sided [-0.08 to 0.05], Standard Error of Mean 0.04 — Mean change calculated as: BI - Placebo
Statistical Analysis 6: Comparison: Placebo Matching to BI 1358894 vs BI 1358894; Mean BOLD signal % change/ Dorsolateral Prefrontal Cortex Right; Test type: Other — [test comment as in outcome 1, analysis 2]; p = 0.8792, ANOVA; Mean change = -0.01, 90% CI 2-sided [-0.09 to 0.07], Standard Error of Mean 0.05 — Mean change calculated as: BI - Placebo
Statistical Analysis 7: Comparison: Placebo Matching to BI 1358894 vs BI 1358894; Mean BOLD signal % change/ Insula Left; Test type: Other — [test comment as in outcome 1, analysis 2]; p = 0.0419, ANOVA; Mean change = -0.08, 90% CI 2-sided [-0.15 to -0.02], Standard Error of Mean 0.04 — Mean change calculated as: BI - Placebo
Statistical Analysis 8: Comparison: Placebo Matching to BI 1358894 vs BI 1358894; Mean BOLD signal % change/ Insula Right; Test type: Other — [test comment as in outcome 1, analysis 2]; p = 0.1658, ANOVA; Mean change = -0.05, 90% CI 2-sided [-0.12 to 0.01], Standard Error of Mean 0.04 — Mean change calculated as: BI - Placebo
Statistical Analysis 9: Comparison: Placebo Matching to BI 1358894 vs Citalopram; Mean BOLD Signal % change/ Amygdala Left; Test type: Other — ANOVA model with treatment (Citalopram versus placebo) and severity of depression (MADRS ≥20 versus <20) as fixed effects. The Citalopram treatment arm was used as a positive control group. It was not planned to compare pharmacodynamic effects between Citalopram and BI 1358894; p = 0.6673, ANOVA; Mean change = -0.02, 90% CI 2-sided [-0.08 to 0.05], Standard Error of Mean 0.04 — Mean change calculated as: BI - Placebo
Statistical Analysis 10: Comparison: Placebo Matching to BI 1358894 vs Citalopram; Mean BOLD Signal % Change/ Amygdala Right; Test type: Other — [test comment as in outcome 1, analysis 9]; p = 0.0778, ANOVA; Mean change = -0.07, 90% CI 2-sided [-0.14 to -0.01], Standard Error of Mean 0.04 — Mean change calculated as: BI - Placebo
Statistical Analysis 11: Comparison: Placebo Matching to BI 1358894 vs Citalopram; Mean BOLD signal % change/ Anterior Cingulate Cortex Left; Test type: Other — [test comment as in outcome 1, analysis 2]; p = 0.3258, ANOVA; Mean change = -0.03, 90% CI 2-sided [-0.08 to 0.02], Standard Error of Mean 0.03 — Mean change calculated as: BI - Placebo
Statistical Analysis 12: Comparison: Placebo Matching to BI 1358894 vs Citalopram; Mean BOLD signal % change/ Anterior Cingulate Cortex Right; Test type: Other — [test comment as in outcome 1, analysis 9]; p = 0.5954, ANOVA; Mean change = -0.02, 90% CI 2-sided [-0.07 to 0.04], Standard Error of Mean 0.03 — Mean change calculated as: BI - Placebo
Statistical Analysis 13: Comparison: Placebo Matching to BI 1358894 vs Citalopram; Mean BOLD signal % change/ Dorsolateral Prefrontal Cortex Left; Test type: Other — [test comment as in outcome 1, analysis 9]; p = 0.5911, ANOVA; Mean change = -0.02, 90% CI 2-sided [-0.08 to 0.04], Standard Error of Mean 0.04 — Mean change calculated as: BI - Placebo
Statistical Analysis 14: Comparison: Placebo Matching to BI 1358894 vs Citalopram; Mean BOLD signal % change/ Dorsolateral Prefrontal Cortex Right; Test type: Other — [test comment as in outcome 1, analysis 9]; p = 0.8283, ANOVA; Mean change = -0.01, 90% CI 2-sided [-0.11 to 0.08], Standard Error of Mean 0.06 — Mean change calculated as: BI - Placebo
Statistical Analysis 15: Comparison: Placebo Matching to BI 1358894 vs Citalopram; Mean BOLD signal % change/ Insula Left; Test type: Other — [test comment as in outcome 1, analysis 9]; p = 0.1797, ANOVA; Mean change = -0.05, 90% CI 2-sided [-0.12 to 0.01], Standard Error of Mean 0.04 — Mean change calculated as: BI - Placebo
Statistical Analysis 16: Comparison: Placebo Matching to BI 1358894 vs Citalopram; Mean BOLD signal % change/ Insula Right; Test type: Other — [test comment as in outcome 1, analysis 9]; p = 0.5772, ANOVA; Mean change = -0.02, 90% CI 2-sided [-0.08 to 0.04], Standard Error of Mean 0.04 — Mean change calculated as: BI - Placebo

2. Secondary Outcome: Mean BOLD Signal % Change in an Emotional Paradigm in the Corticolimbic System Using the Affective Pictures of the Open Affective Standardised Image Set (OASIS).
Description: The secondary endpoint was the mean BOLD signal % change in an emotional paradigm (affective picture set - OASIS task) in the corticolimbic system, consisting of eight brain regions:
  * Amygdala left
  * Amygdala right
  * Dorsolateral prefrontal cortex left
  * Dorsolateral prefrontal cortex right
  * Insula left
  * Insula right
  * Anterior cingulate cortex left
  * Anterior cingulate cortex right
Time Frame: A 50 min scan, 6 hours following drug intake.
Population: Evaluable set (ES): This patient set included all randomised patients who performed the fMRI measurements and did not experience severe headaches directly before or during the fMRI measurements. In particular, patients who had to be replaced due to severe headaches were excluded from the ES.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Placebo Matching to BI 1358894 | Citalopram | BI 1358894
Number analyzed (Participants) | 24 | 23 | 22
Percent change
  Amygdala left | 0.231 (0.123) | 0.185 (0.130) | 0.148 (0.100)
  Amygdala right | 0.200 (0.125) | 0.186 (0.130) | 0.132 (0.105)
  Dorsolateral prefrontal cortex left | 0.269 (0.132) | 0.262 (0.178) | 0.147 (0.141)
  Dorsolateral prefrontal cortex right | 0.229 (0.174) | 0.220 (0.116) | 0.155 (0.141)
  Insula left | 0.279 (0.132) | 0.270 (0.125) | 0.164 (0.114)
  Insula right | 0.195 (0.142) | 0.207 (0.154) | 0.120 (0.100)
  Anterior cingulate cortex left | 0.089 (0.100) | 0.071 (0.081) | 0.027 (0.110)
  Anterior cingulate cortex right | 0.091 (0.129) | 0.082 (0.113) | 0.025 (0.104)
Statistical Analysis 1: Comparison: Placebo Matching to BI 1358894 vs BI 1358894; Mean BOLD signal % change/ Amygdala Left; Test type: Other — [test comment as in outcome 1, analysis 2]; p = 0.0147, ANOVA; Mean change = -0.09, 90% CI 2-sided [-0.14 to -0.03], Standard Error of Mean 0.03 — Mean change calculated as: BI - Placebo
Statistical Analysis 2: Comparison: Placebo Matching to BI 1358894 vs BI 1358894; Mean BOLD signal % change/ Amygdala Right; Test type: Other — [test comment as in outcome 1, analysis 2]; p = 0.0480, ANOVA; Mean change = -0.07, 90% CI 2-sided [-0.13 to -0.01], Standard Error of Mean 0.03 — Mean change calculated as: BI - Placebo
Statistical Analysis 3: Comparison: Placebo Matching to BI 1358894 vs BI 1358894; Mean BOLD signal % change/ Anterior Cingulate Cortex Left; Test type: Other — [test comment as in outcome 1, analysis 2]; p = 0.0294, ANOVA; Mean change = -0.07, 90% CI 2-sided [-0.12 to -0.02], Standard Error of Mean 0.03 — Mean change calculated as: BI - Placebo
Statistical Analysis 4: Comparison: Placebo Matching to BI 1358894 vs BI 1358894; Mean BOLD signal % change/ Anterior Cingulate Cortex Right; Test type: Other — [test comment as in outcome 1, analysis 2]; p = 0.0359, ANOVA; Mean change = -0.07, 90% CI 2-sided [-0.13 to -0.02], Standard Error of Mean 0.03 — Mean change calculated as: BI - Placebo
Statistical Analysis 5: Comparison: Placebo Matching to BI 1358894 vs BI 1358894; Mean BOLD signal % change/ Dorsolateral Prefrontal Cortex Left; Test type: Other — [test comment as in outcome 1, analysis 2]; p = 0.0022, ANOVA; Mean change = -0.13, 90% CI 2-sided [-0.19 to -0.06], Standard Error of Mean 0.04 — Mean change calculated as: BI - Placebo
Statistical Analysis 6: Comparison: Placebo Matching to BI 1358894 vs BI 1358894; Mean BOLD signal % change/ Dorsolateral Prefrontal Cortex Right; Test type: Other — [test comment as in outcome 1, analysis 2]; p = 0.1040, ANOVA; Mean change = -0.08, 90% CI 2-sided [-0.15 to 0.00], Standard Error of Mean 0.05 — Mean change calculated as: BI - Placebo
Statistical Analysis 7: Comparison: Placebo Matching to BI 1358894 vs BI 1358894; Mean BOLD signal % change/ Insula Left; Test type: Other — [test comment as in outcome 1, analysis 2]; p = 0.0022, ANOVA; Mean change = -0.12, 90% CI 2-sided [-0.18 to -0.06], Standard Error of Mean 0.04 — Mean change calculated as: BI - Placebo
Statistical Analysis 8: Comparison: Placebo Matching to BI 1358894 vs BI 1358894; Mean BOLD signal % change/ Insula Right; Test type: Other — [test comment as in outcome 1, analysis 2]; p = 0.0331, ANOVA; Mean change = -0.08, 90% CI 2-sided [-0.14 to -0.02], Standard Error of Mean 0.04 — Mean change calculated as: BI - Placebo
Statistical Analysis 9: Comparison: Placebo Matching to BI 1358894 vs Citalopram; Mean BOLD signal % change/ Amygdala Left; Test type: Other — [test comment as in outcome 1, analysis 9]; p = 0.2149, ANOVA; Mean change = -0.05, 90% CI 2-sided [-0.11 to 0.02], Standard Error of Mean 0.04 — Mean change calculated as: BI - Placebo
Statistical Analysis 10: Comparison: Placebo Matching to BI 1358894 vs Citalopram; Mean BOLD signal % change/ Amygdala Right; Test type: Other — [test comment as in outcome 1, analysis 9]; p = 0.6896, ANOVA; Mean change = -0.02, 90% CI 2-sided [-0.08 to 0.05], Standard Error of Mean 0.04 — Mean change calculated as: BI - Placebo
Statistical Analysis 11: Comparison: Placebo Matching to BI 1358894 vs Citalopram; Mean BOLD signal % change/ Anterior Cingulate Cortex Left; Test type: Other — [test comment as in outcome 1, analysis 9]; p = 0.4769, ANOVA; Mean change = -0.02, 90% CI 2-sided [-0.06 to 0.02], Standard Error of Mean 0.03 — Mean change calculated as: BI - Placebo
Statistical Analysis 12: Comparison: Placebo Matching to BI 1358894 vs Citalopram; Mean BOLD signal % change/ Anterior Cingulate Cortex Right; Test type: Other — [test comment as in outcome 1, analysis 9]; p = 0.7680, ANOVA; Mean change = -0.01, 90% CI 2-sided [-0.07 to 0.05], Standard Error of Mean 0.03 — Mean change calculated as: BI - Placebo
Statistical Analysis 13: Comparison: Placebo Matching to BI 1358894 vs Citalopram; Mean BOLD signal % change/ Dorsolateral Prefrontal Cortex Left; Test type: Other — [test comment as in outcome 1, analysis 2]; p = 0.7997, ANOVA; Mean change = -0.01, 90% CI 2-sided [-0.08 to 0.06], Standard Error of Mean 0.04 — Mean change calculated as: BI - Placebo
Statistical Analysis 14: Comparison: Placebo Matching to BI 1358894 vs Citalopram; Mean BOLD signal % change/ Dorsolateral Prefrontal Cortex Right; Test type: Other — [test comment as in outcome 1, analysis 9]; p = 0.8334, ANOVA; Mean change = -0.01, 90% CI 2-sided [-0.08 to 0.06], Standard Error of Mean 0.04 — Mean change calculated as: BI - Placebo
Statistical Analysis 15: Comparison: Placebo Matching to BI 1358894 vs Citalopram; Mean BOLD signal % change/ Insula Left; Test type: Other — [test comment as in outcome 1, analysis 9]; p = 0.7402, ANOVA; Mean change = -0.01, 90% CI 2-sided [-0.07 to 0.05], Standard Error of Mean 0.04 — Mean change calculated as: BI - Placebo
Statistical Analysis 16: Comparison: Placebo Matching to BI 1358894 vs Citalopram; Mean BOLD signal % change/ Insula Right; Test type: Other — [test comment as in outcome 1, analysis 9]; p = 0.8120, ANOVA; Mean change = 0.01, 90% CI 2-sided [-0.06 to 0.08], Standard Error of Mean 0.04 — Mean change calculated as: BI - Placebo

ADVERSE EVENTS:
Time Frame: From the time of administration of BI 1358894 or BI-matching placebo (in the placebo and Citalopram arm) until time of administration of BI 1358894 or BI-matching placebo + Residual effect period(14*24 h) or 0:00 AM on day after subject's trial termination date, whatever occurs earlier. Up to 14 days.
Description: Safety Set (SS): This subject set includes all randomised patients who received the study drugs (BI 1358894, Citalopram or placebo). Patient randomized to the BI 1358894 but received Placebo at both time points.
Groups:
- BI 1358894 +Citalopram: This column is based on the treatment the patients actually did receive.
  Patient randomized to the Citalopram but received BI 1358894 instead of Placebo at the first planned time point.
  Citalopram blood concentrations of patient, randomised to BI 1358894, showed that the Patient has received but did not report Citalopram as co-medication, at an unknown dose.
Arm/Group | Placebo Matching to BI 1358894 | Citalopram | BI 1358894 | BI 1358894 +Citalopram
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/23 | 0/23 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/23 | 0/23 | 0/2
Other Adverse Events (participants affected / at risk) | 13/25 | 13/23 | 21/23 | 2/2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Matching to BI 1358894 (N=25) | Citalopram (N=23) | BI 1358894 (N=23) | BI 1358894 +Citalopram (N=2)
Headache (Nervous system disorders) | 10 | 12 | 17 | 1
Dizziness (Nervous system disorders) | 1 | 1 | 3 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 1 | 0 | 1
Fatigue (General disorders) | 0 | 4 | 4 | 0
Nasopharyngitis (Infections and infestations) | 2 | 0 | 3 | 0
Nausea (Gastrointestinal disorders) | 3 | 1 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2019-02-21): https://cdn.clinicaltrials.gov/large-docs/78/NCT03854578/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-22): https://cdn.clinicaltrials.gov/large-docs/78/NCT03854578/SAP_001.pdf